CLINICAL TRIAL: NCT03965468
Title: A Multicentre Single Arm Phase II Trial Assessing the Efficacy of Immunotherapy, Chemotherapy and Stereotactic Radiotherapy to Metastases Followed by Definitive Surgery or Radiotherapy to the Primary Tumour, in Patients With Synchronous Oligo-metastatic Non-small Cell Lung Cancer
Brief Title: Immunotherapy, Chemotherapy, Radiotherapy and Surgery for Synchronous Oligo-metastatic NSCLC
Acronym: CHESS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 14-18; 2018-003011-22 (EudraCT Number); ESR-17-13224 (Other: AstraZeneca)
Record Dates: First submitted 2019-05-24; First posted 2019-05-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer; Stage IV; Oligometastasis
Keywords: NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab; Carboplatin; Paclitaxel; Radiosurgery; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immunotherapy, chemotherapy, radiotherapy and surgery (Experimental): Durvalumab 1500 mg administered intravenously every 3 weeks for the first 4-6 cycles (during chemotherapy);
  Tremelimumab 75mg administered intravenously every 3 weeks for the first 4-6 cycles (only cohort 2)
  4-6 cycles of chemotherapy, carboplatin AUC5 every 3 weeks plus paclitaxel 175 mg/m2, every 3 weeks;
  Stereotactic body radiotherapy (SBRT) of all oligo-metastatic lesions, in a maximum of 10 treatment fractions over 2 weeks, starting after week one of chemotherapy cycle 1 and completed within four weeks after start of durvalumab treatment;
  Restaging at 3 months; if no disease progression, proceed to definitive local treatment (surgical resection of primary tumour or radiotherapy at a minimum dose of 60-66Gy to the primary tumour). Durvalumab continues at 1500 mg intravenously every 4 weeks until progression of disease or for a maximum of 1 year from start of treatment.
  Interventions: Drug: Durvalumab; Drug: Carboplatin; Drug: Paclitaxel; Radiation: Stereotactic body radiation therapy (SBRT); Procedure: Surgical resection - definitive local treatment.; Radiation: Radical radiotherapy - definitive local treatment.; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is a human monoclonal antibody (mAb) of the immunoglobulin G (IgG) 1 kappa subclass that inhibits binding of PD-L1. Durvalumab is expected to stimulate the patient's antitumour immune response by binding to PD L1 and shifting the balance toward an antitumour response.
  Other Names: Imfinzi
Drug: Carboplatin — Carboplatin belongs to the group of medicines known as alkylating agents. Carboplatin interferes with the growth of cancer cells, which eventually are destroyed.
Drug: Paclitaxel — A compound extracted from the Pacific yew tree Taxus brevifolia with antineoplastic activity. Paclitaxel binds to tubulin and inhibits the disassembly of microtubules, thereby resulting in the inhibition of cell division. This agent also induces apoptosis by binding to and blocking the function of the apoptosis inhibitor protein Bcl-2 (B-cell Leukemia 2).
Radiation: Stereotactic body radiation therapy (SBRT) — SBRT of all oligo-metastatic lesions
Procedure: Surgical resection - definitive local treatment. — Surgical resection of primary tumour for patients with single station, non-bulky tumours.
Radiation: Radical radiotherapy - definitive local treatment. — Conventional or moderately hypo-fractionated radiotherapy to the primary tumour for other tumour stages, or in case of medical inoperability.
Drug: Tremelimumab — Tremelimumab is a human mAb of the IgG 2 subclass that is directed against CTLA-4 (CD152), a cell surface receptor that is expressed primarily on activated T-cells and acts to inhibit their activation. Tremelimumab completely blocks the interaction of human CTLA-4 with CD80 and CD86, resulting in increased release of cytokines (interleukin-2 and IFN-γ) from human T-cells, peripheral blood mononuclear cells and whole blood.

SUMMARY:
A multicentre single arm phase II trial assessing the efficacy of immunotherapy, chemotherapy plus stereotactic radiotherapy to metastases followed by definitive surgery or radiotherapy to the locoregional primary tumour, in patients with histologically-confirmed synchronous oligo-metastatic non-small cell lung cancer (NSCLC).

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) continues to be the leading cause of cancer-related mortality worldwide. Even with adjustment for age NSCLC is responsible for almost 20% of cancer-related deaths. Recent years have brought tremendous progress in the understanding of the disease, its underlying biology and the development of effective therapies. Traditionally, NSCLC has been treated with surgery, platinum-based chemotherapy or radiotherapy alone or in combination, depending on tumour stage, tolerability of expected side effects and prognosis. Various strategies are currently being pursued in order to increase the patient population that may benefit from immunotherapy and to further improve the outcome of patients with NSCLC.

The CHESS clinical trial is for patients with NSCLC that has progressed to a small number of other parts of the body (oligo-metastatic) and has not been previously treated, or after surgical resection of a single metastasis (central nervous system or adrenal). The trial aims to reduce the risk of systemic progression and thereby improve progression free survival. Participants will receive induction treatment consisting of immunotherapy combined with platinum-based doublet chemotherapy and stereotactic body radiotherapy (SBRT) that will be given to all oligo-metastatic locations. SBRT started early and concurrently with immunotherapy aims at enhancing a postulated immune effect and simultaneously effectively control the macro-metastases.

Preclinical data have shown a strong immune-enhancing effect of radiotherapy, especially when delivered to small volumes, in high-single fraction doses and over a short period of time. Consequently, stereotactic body radiotherapy (SBRT) is currently being intensively investigated as a partner for systemic immunotherapy. Earlier clinical studies generated proof-of-principle data for the synergistic effects of combined radiotherapy and immunotherapy. Chemotherapy and high-dose radiotherapy are well known triggers of immunogenic cell death and are therefore highly promising partners for combination with immunotherapy.

The sub-group of patients with "oligometastatic" disease was originally described by Hellman and Weichselbaum in 1995. In line with this concept, the current NCCN and ESMO guidelines describe that Stage IV NSCLC patients presenting with solitary metastases can be treated with curative intent using local surgery and/or radiotherapy. Local treatment for oligo-metastatic NSCLC has been adopted rapidly in the oncological community and one reason is the progress made in the fields of surgery and radiotherapy, both becoming less toxic (minimally invasive surgery) and simultaneously less toxic and more effective (precision radiotherapy), respectively. SBRT allows treatment of small peripheral primaries and metastases at virtually all anatomical locations with a favourable therapeutic ratio of local tumour control rates >90% and low rates of toxicity. Simultaneously, minimally invasive surgery for early and locally advanced NSCLC today achieves excellent local tumour control with low rates of toxicity.

Patients with a limited number of metastases - oligometastatic disease - are currently treated with combined radical local treatment for all active lesions (locoregional primary and metastases) and their prognosis is better as compared to patients who receive systemic treatment only for widespread metastatic disease. However, the majority of patients still develop systemic disease progression indicating the urgent clinical need for more effective systemic treatment to control subclinical disease.

All CHESS trial participants will receive induction treatment with the immunotherapy drug durvalumab, standard platinum-chemotherapy and radiation therapy of the lung cancer metastases (SBRT). Durvalumab is a human monoclonal antibody carefully engineered to attach to immune cells to stimulate their activity against cancer cells. There are now several approved antibodies for the treatment of cancer or other diseases. Standard platinum-chemotherapy includes treatment with carboplatin and paclitaxel.

After three months of induction treatment the status of the lung cancer will be restaged. If the primary lung cancer is stable or has not increased in size it will be surgically removed if possible or, alternatively, treated with radiation therapy. Treatment with durvalumab will continue until the disease relapses or for a maximum of one year from the start of induction treatment. If the lung cancer has increased in size at the time of the three month restaging all trial treatment will stop and the study doctor will discuss other treatment options that are available.

The efficacy, safety and tolerability of combining immunotherapy with standard platinum-chemotherapy and SBRT will be evaluated in the CHESS clinical trial.

Encouraged by the positive results of the POSEIDON trial, we amended the CHESS protocol to include a second cohort of additional 47 patients who will receive tremelimumab, in addition to the protocol treatment of the original CHESS protocol (e.g., durvalumab, platinum-based doublet chemotherapy, and SRBT to the oligo-metastatic lesions, followed by definitive local treatment for patients that have not progressed at the time of restaging).

Objectives and endpoints, patient selection and statistical assumption remain the same as for cohort 1 in the original protocol.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed non-small cell lung cancer
* Synchronous oligo-metastatic stage IV disease: maximum of three distant metastases, one of which must be extra-cerebral for stereotactic body radiotherapy (SBRT); Initial mediastinal staging is recommended (except for lymph nodes <1 cm on CT and PET-negative) preferentially by endobronchial ultrasound (EBUS); Neurosurgical resection of one single central nervous system (CNS) metastasis or laparoscopic resection of one adrenal metastasis before study inclusion is allowed (one extra-cerebral metastasis must be available for SBRT)
* Able to understand and give written informed consent and comply with study procedures
* Age ≥18 years
* ECOG Performance Status 0-1
* Availability of tumour tissue for translational research
* Adequate haematological, renal and liver function

Exclusion Criteria:

* Prior chemotherapy, radiotherapy or therapeutic surgery for NSCLC (an exception is the resection of one single CNS or adrenal metastasis, as above)
* Activating driver mutation: epidermal growth factor receptor (EGFR), anaplastic lymphoma kinase (ALK), proto-oncogene receptor tyrosine kinase (ROS1)
* More than three distant metastases
* Brain metastases not amendable for radiosurgery or neurosurgery
* Extracranial metastatic locations such as malignant ascites, pleural or pericardial effusion, diffuse lymphangiomatosis of skin or lung, diffuse bone marrow metastasis, abdominal masses/abdominal organomegaly, identified by physical exam that is not measurable by reproducible imaging techniques.
* Primary lung cancer not suitable for radical therapy (pneumonectomy excluded)
* History of leptomeningeal carcinomatosis
* Major surgery or significant traumatic injury from which the patient has not recovered at least 28 days before enrolment
* Any uncontrolled intercurrent illness, including but not limited to: ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease or serious chronic gastrointestinal conditions associated with diarrhea, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol
* Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc) at screening.
* Known positivity for human immunodeficiency virus (positive HIV 1/2 antibodies) or active tuberculosis infection (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice)
* Active autoimmune disease requiring systemic treatment
* Severe or uncontrolled cardiac disease requiring treatment
* History of active primary immunodeficiency
* History of allogeneic organ transplant
* Receipt of live attenuated vaccines within 30 days prior to enrolment
* Known allergies or hypersensitivity to trial drugs or to any excipient.
* Women who are pregnant or in the period of lactation.
* Sexually active men and women of childbearing potential who are not willing to use a highly effective contraceptive method during the trial and up to 90 days after last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab and tremelimumab combination therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2019-11-19 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival at 12 months | Assessed from the date of enrolment to completion of treatment at 12 months.
  The PFS rate at 1-year is the primary endpoint of this trial and it is defined as the rate of patients without a PFS event at 1-year after enrolment. The rate will be estimated as the percentage of patients without a PFS event over the total number of patients who have completed a 1-year follow-up period after the enrolment. PFS is defined as the time from the date of enrolment until documented progression or death, if progression is not documented. Progression is defined as the development of new metastatic lesions or local progression of resected or irradiated metastases or primary tumour, assessed according to RECIST criteria version 1.1

SECONDARY OUTCOMES:
Overall survival | Time from date of enrolment until death from any cause. Assessed for up to 30 months.
  Overall survival (OS) is defined as the time from the date of enrolment until death from any cause. Censoring for OS (patients without reported death) will occur at the last follow-up date.
Pattern of disease progression | Assessed from the date of enrolment until progression, from enrolment up to 12 months.
  Defined as the site of first progression. None, locoregional, distant, or both locoregional and distant.
Response to induction therapy | Assessed from the start of protocol treatment until the 3-month restaging
  Defined as the best overall response [complete response (CR) or partial response (PR)] according to RECIST 1.1 criteria.
Distant progression-free survival | Assessed from the date of enrolment for up to 12 months.
  Defined as the date of development of new metastases, excluding oligometastasis diagnosed at enrolment.
Overall response | Assessed from the start of protocol treatment across all time points until the end of follow-up, assessed for up to 30 months.
  Defined as best overall response [complete response (CR) or partial response (PR) according to RECIST 1.1 criteria.
Duration of response | Assessed from the date of enrolment for up to 12 months.
  Defined as the interval from the date of first documentation of objective response (CR or PR), according to RECIST 1.1 criteria to the date of first documented progression, relapse or death from any cause.
Symptom-specific and global quality of life: The Lung Cancer Symptom Scale | Assessed at trial entry, until 6 months after treatment start and at 12 months from enrolment.
  The Lung Cancer Symptom Scale, a 9-item one page questionnaire will be used to assess change in total score (average of all 9 items).
Toxicity before and after surgery/radiotherapy | Adverse events will be collected from the date of consent until 90 days after the completion of treatment.
  Safety parameters will be assessed in terms of adverse events graded by CTCAE v5.0 including events leading to dose interruptions, withdrawals of protocol treatment and death; severe, serious and selected adverse events; deaths; clinically significant laboratory parameters and abnormalities, and vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, MD-PhD, Study Chair — University Hospital, Zürich; Isabelle Schmitt-Opitz, MD, Study Chair — University Hospital, Zürich
Locations (15):
- Italy (3):
  - European Institute of Oncology, Milan
  - Istituto Oncologico Veneto - Irccs, Padua
  - IRCCS Istituto Nazionale Tumori Regina Elena, Roma
- Netherlands (2):
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medical Centre, Rotterdam
- Spain (5):
  - Hosp. De la Santa Creu i Sant Pau, Barcelona
  - Hosp. Uni. Virgen de las Nieves, Granada
  - Hosp. Sanchinarro- Centro Integral Oncología Clara Campal, Madrid
  - Vall d'Hebron University Hospital, Madrid
  - Hosp. Uni. Politécnico La Fe, Valencia
- Switzerland (5):
  - Inselspital Bern, Bern
  - Geneva University Hospital, Geneva
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Kantonsspital Winterthur, Winterthur
  - University Hospital Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Galluzzi L, Buque A, Kepp O, Zitvogel L, Kroemer G. Immunogenic cell death in cancer and infectious disease. Nat Rev Immunol. 2017 Feb;17(2):97-111. doi: 10.1038/nri.2016.107. Epub 2016 Oct 17. PMID 27748397
- [Background] Langer CJ, Gadgeel SM, Borghaei H, Papadimitrakopoulou VA, Patnaik A, Powell SF, Gentzler RD, Martins RG, Stevenson JP, Jalal SI, Panwalkar A, Yang JC, Gubens M, Sequist LV, Awad MM, Fiore J, Ge Y, Raftopoulos H, Gandhi L; KEYNOTE-021 investigators. Carboplatin and pemetrexed with or without pembrolizumab for advanced, non-squamous non-small-cell lung cancer: a randomised, phase 2 cohort of the open-label KEYNOTE-021 study. Lancet Oncol. 2016 Nov;17(11):1497-1508. doi: 10.1016/S1470-2045(16)30498-3. Epub 2016 Oct 10. PMID 27745820
- [Background] Rizvi NA, Hellmann MD, Brahmer JR, Juergens RA, Borghaei H, Gettinger S, Chow LQ, Gerber DE, Laurie SA, Goldman JW, Shepherd FA, Chen AC, Shen Y, Nathan FE, Harbison CT, Antonia S. Nivolumab in Combination With Platinum-Based Doublet Chemotherapy for First-Line Treatment of Advanced Non-Small-Cell Lung Cancer. J Clin Oncol. 2016 Sep 1;34(25):2969-79. doi: 10.1200/JCO.2016.66.9861. Epub 2016 Jun 27. PMID 27354481
- [Background] Twyman-Saint Victor C, Rech AJ, Maity A, Rengan R, Pauken KE, Stelekati E, Benci JL, Xu B, Dada H, Odorizzi PM, Herati RS, Mansfield KD, Patsch D, Amaravadi RK, Schuchter LM, Ishwaran H, Mick R, Pryma DA, Xu X, Feldman MD, Gangadhar TC, Hahn SM, Wherry EJ, Vonderheide RH, Minn AJ. Radiation and dual checkpoint blockade activate non-redundant immune mechanisms in cancer. Nature. 2015 Apr 16;520(7547):373-7. doi: 10.1038/nature14292. Epub 2015 Mar 9. PMID 25754329
- [Background] Kang J, Demaria S, Formenti S. Current clinical trials testing the combination of immunotherapy with radiotherapy. J Immunother Cancer. 2016 Sep 20;4:51. doi: 10.1186/s40425-016-0156-7. eCollection 2016. PMID 27660705
- [Background] Bernstein MB, Krishnan S, Hodge JW, Chang JY. Immunotherapy and stereotactic ablative radiotherapy (ISABR): a curative approach? Nat Rev Clin Oncol. 2016 Aug;13(8):516-24. doi: 10.1038/nrclinonc.2016.30. Epub 2016 Mar 8. PMID 26951040
- [Background] Golden EB, Chhabra A, Chachoua A, Adams S, Donach M, Fenton-Kerimian M, Friedman K, Ponzo F, Babb JS, Goldberg J, Demaria S, Formenti SC. Local radiotherapy and granulocyte-macrophage colony-stimulating factor to generate abscopal responses in patients with metastatic solid tumours: a proof-of-principle trial. Lancet Oncol. 2015 Jul;16(7):795-803. doi: 10.1016/S1470-2045(15)00054-6. Epub 2015 Jun 18. PMID 26095785
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Weichselbaum RR, Hellman S. Oligometastases revisited. Nat Rev Clin Oncol. 2011 Jun;8(6):378-82. doi: 10.1038/nrclinonc.2011.44. Epub 2011 Mar 22. PMID 21423255